CLINICAL TRIAL: NCT01817231
Title: Vitamin D Status and Breast Cancer in Saudi Arabian Women: Case Control Study
Brief Title: Epidemiological Analysis of Vitamin D and Breast Cancer Risk in Saudi Arabian Women
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Cynthia Thomson, Professor College of Public Health, University of Arizona
Other Study IDs: SAVitaminD
Record Dates: First submitted 2013-03-12; First posted 2013-03-25 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer; Vitamin D Deficiency
Keywords: breast cancer; vitamin D; 25 OH vitamin D
MeSH Terms: conditions — Breast Neoplasms; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum for vitamin D levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- breast cancer cases: breast cancer cases versus controls

SUMMARY:
This is an analysis of de-identified data collected from 240 Saudi Arabian women, 120 with breast cancer and 120 control women, to evalyate if vitamin D status is associated with breast cancer risk.

DETAILED DESCRIPTION:
Background: The role of vitamin D in breast cancer prevention is equivocal. Saudi Arabian women are thought to be at greater risk for vitamin D deficiency due to darker skin type and greater likelihood for reduced UVB radiation exposure. However, there is a lack of data regarding the vitamin D status of Saudi Arabian women and how this may relate to breast cancer risk.

Objective: The purpose of this research was to evaluate the association between circulating concentrations of 25(OH)D and breast cancer risk in Saudi Arabian women.

Design: A case-control study was conducted among 120 breast cancer cases and 120 controls. The study population was drawn from patients admitted to King Fahd Hospital in Jeddah, Saudi Arabia from June to August 2009. Participants completed questionnaires on diet and medical history and serum samples were collected from all women to measure circulating 25(OH)D concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer (cases) or healthy women (controls),
* receiving standard medical check-ups at the women's clinic
* Female,
* between the ages of 18 and 75 years
* BMI ≤ 40 kg/m2
* residence in Saudi Arabia for more than 5 years
* absence of chronic diseases that could affect vitamin D metabolism, including renal, hepatic, endocrine, or autoimmune disease.

Exclusion Criteria:

receiving standard medical check-ups at the women's clinic

* Male,
* less than 18 or greater than 75 years of age
* BMI > 40 kg/m2
* Not a resident of Saudi Arabia for more than 5 years
* Presence of chronic diseases that could affect vitamin D metabolism, including renal, hepatic, endocrine, or autoimmune disease.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Saudi Arabian women receiving care at King Fahd Women's clinic in Saudi Arabia during the summer of 2009.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
serum vitamin D | cross-sectional from May 2009-August 2009
  assessed serum vitamin D in cases versus controls

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Thomson, PhD, Study Chair — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Derived] Yousef FM, Jacobs ET, Kang PT, Hakim IA, Going S, Yousef JM, Al-Raddadi RM, Kumosani TA, Thomson CA. Vitamin D status and breast cancer in Saudi Arabian women: case-control study. Am J Clin Nutr. 2013 Jul;98(1):105-10. doi: 10.3945/ajcn.112.054445. Epub 2013 May 22. PMID 23697705